CLINICAL TRIAL: NCT01765374
Title: Study of Sonographic Efficacy of Rituximab in Rheumatoid Arthritis
Acronym: SEWORRA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2010/081/HP
Record Dates: First submitted 2011-05-12; First posted 2013-01-10 (Estimated); Last update posted 2015-01-22 (Estimated); Status verified 2015-01

CONDITIONS: Rheumatoid Arthritis
Keywords: rituximab; sonography; clinical response
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Ultrasonography; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- rituximab (Experimental): Only one arm; all patients are treated by rituximab (monotherapy or in combination with conventional DMARD)
  Interventions: Device: ESAOTE MyLab60; Drug: Rituximab

INTERVENTIONS:
Device: ESAOTE MyLab60 — US evaluation at different time points
  Other Names: sonography
Drug: Rituximab

SUMMARY:
To detect by sonography relapse of disease activity prior to clinical symptoms in RA patients treated by rituximab.

ELIGIBILITY:
Inclusion Criteria:

* failure to at least one TNF-blocking agent

Exclusion Criteria:

* pregnant or childbearing woman
* Rituximab contraindication
* woman unable to use contraceptive means

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2011-02; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
global score of power-doppler activity measured by ultrasonography on 12 joints | at 6 months after initiation of rituximab and then every 2 month over the follow-up period (18 months)
  Each time point will be assessed since the main objective of the study is to detect the time of sonographic relapse prior to clinical relapse

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Vittecoq, MD,PHD, Principal Investigator — University Hospital, Rouen
Locations (5):
- France (5):
  - Department of Rheumatology, CHU de Caen, Caen
  - Normandy, Caen, Le Havre, Rouen, Elbeuf
  - Department of Rheumatology, Le Havre
  - Department of rheumatology, Rouen
  - Department of Rheumatology CHG Elbeuf, Saint-Aubin-lès-Elbeuf